CLINICAL TRIAL: NCT04884425
Title: A Pilot Randomised Controlled Feasibility Trial for the Use of a Pulsed Electromagnetic Field Device to Assist Management of Type 2 Diabetes
Brief Title: A Trial for the Use of a Pulsed Electromagnetic Field Device to Assist Management of Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St Mary's University College (Other)
Collaborators: Energy5 Limited (Unknown)
Responsible Party: Principal Investigator, Anne Majumdar, Research Administrator, St Mary's University College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SMU_ETHICS_2020-21_157
Record Dates: First submitted 2021-05-04; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Type 2 Diabetes
Keywords: Pulsed Electromagnetic Frequency Device; Diabetic Pain
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Consenting participants will be randomised into either the PEMF device group or the waiting list control group. There will be 30 participants in the PEMF group and 30 in the waiting list control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEMF Device Group (Active Comparator): This arm will consist of participant's who have been randomly assigned to use the PEMF device daily for 30 mins for an overall 3 months
  Interventions: Device: Pulsed Electromagnetic Frequency Device (Energy5)
- Waiting List Control Group (No Intervention): These participants will be randomly selected to be on the waiting list group. All waiting list participants will be offered the use of the PEMF device after the study has completed

INTERVENTIONS:
Device: Pulsed Electromagnetic Frequency Device (Energy5) — A pulsed electromagnetic frequency (PEMF) device which is recommended to be used for 30 minutes a day
  Other Names: Energy5
  Arms: PEMF Device Group

SUMMARY:
The majority of people with diabetes worldwide consist of type 2 diabetes mellitus. Typically, patients with type 2 diabetes are encouraged to manage their condition with weight loss; healthy eating; regular exercise; blood glucose monitoring; and in some cases, diabetes medication or insulin therapy. However, many struggle with their condition.

Pulsed Electromagnetic Frequency (PEMF) devices, which follow similar principles as a TENS machine, emit electromagnetic fields and are proposed to provide a non-invasive, safe, and easy-to-use method for treatment and management of diabetes related symptoms such as pain, alongside existing treatments and interventions. There is a belief that such devices may promote health and wellbeing and as a result could improve outcomes of type 2 diabetes. The use of the PEMF device would not replace existing treatments, interventions, or any primary care that the participants are currently receiving.

The purpose of this study is to evaluate the effectiveness of a PEMF device of this kind for reported symptoms such as pain, fatigue, and overall wellbeing in people with type 2 diabetes. The study also seeks to explore patients' experiences of using the PEMF device.

DETAILED DESCRIPTION:
Type 2 diabetes is highly prevalent and many sufferers struggle with their condition. One symptom of type 2 diabetes is diabetic neuropathy, which is characterised by progressive pain and loss of sensation.

Pulsed Electromagnetic Frequency (PEMF) devices, which follow similar principles as a TENS machine, emit electromagnetic fields and are proposed to provide a non-invasive, safe, and easy-to-use method for treatment and management of pain alongside existing treatments and interventions. A recent systematic review reported that pulsed electromagnetic fields had high efficacy in reducing musculoskeletal pain and that methods were well tolerated and had no negative side effects. Research established that pulsed electromagnetic field therapy had beneficial effects on pain, stiffness, and physical function in patients with osteoarthritis. It has, however, been recommended that further research is conducted to examine the use and effectiveness of pulsed electromagnetic field methods.

Given the findings reported regarding the effectiveness of pulsed electromagnetic field methods in reducing pain, it is possible that such devices could prove effective in managing diabetes related symptoms such as pain. It would also be useful to provide insight on the claim that they could potentially improve outcomes of type 2 diabetes and benefit users overall wellbeing.

The study is a pragmatic study as it is considered a better reflection of the perceived clinical benefits in a real world setting as opposed to being more efficacious in a trial setting. Pragmatic studies answer questions such as whether there is perceived additional clinical benefit where a treatment is utilised alongside usual care. This can then determine whether there is reason to explore this matter further and conduct a placebo-controlled trial to further inform health professionals and clinical guidelines.

The purpose of this study, therefore, is to evaluate the effectiveness of a pulsed electromagnetic field (PEMF) device for managing pain, health and wellbeing issues associated with type 2 diabetes via a pragmatic study. The study also seeks to explore patients' experiences of using the device.

Objectives:

1. To evaluate the effectiveness of the PEMF device for symptoms associated with type 2 diabetes.
2. To evaluate the effectiveness of the PEMF device for quality of life in patients with type 2 diabetes.
3. To explore type 2 diabetes patients' experiences of using the PEMF device.

This is a mixed methods study containing quantitative questionnaires and some qualitative interviews. All methods are non-evasive. The target population will be a heterogeneous and demographically diverse group of patients with type 2 diabetes meeting the inclusion criteria. Patients will be aged 18 years and over with a diagnosis of type 2 diabetes. Patients must be willing to participate, be able to read and write in English, and be able to give full, informed, written consent.

Patients will be recruited from patient support groups for adults with type 2 diabetes. In addition, the screening process will exclude those ineligible for inclusion. Responses to an on-line link will highlight the particulars of those interested in participating. Research staff will email an invitation letter to selected respondents (as per the study inclusion criteria ) with type 2 diabetes, together with a screening questionnaire, a patient information sheet and a consent form. Those who indicate they are interested in participating will be further contacted by the research team.

Consenting participants will be randomised into either the PEMF device group or the waiting list control group. There will be 30 participants in the PEMF group and 30 in the waiting list control group. The trial period of device use will last 3 months. Participants will be asked to use the PEMF device for 30 minutes per day.

The study outcome measures will assess diabetes symptoms and quality of life, and will be completed at baseline and at the end of the study intervention. All questionnaire tools have been previously validated. The Interview schedule will be piloted prior to use. Outcome measures consist of the following validated instruments: the Appraisal of Diabetes Scale (ADS), Measure Yourself Medical Outcome Profile (MYMOP)2, and the EQ-5D-5L tool to determine health related quality of life.The outcome measures will be collected at baseline, 6-weeks, 3 months plus a 6 month follow up.

Participants will be asked to complete a patient diary throughout the duration of the trial. The diary will ask participants to indicate use of study interventions, use of prescribed and non-prescribed treatments, and use of NHS services during the course of the trial. The diary will additionally record details of any changes to participants' food consumption during the trial period, device usage, and any routine blood glucose monitoring.

Sociodemographic and treatment characteristics will be obtained from a participants demographics questionnaire. These will include gender, age, educational level, marital status, and diabetes treatment received and dosage.

Participants will be invited to send the study team any clinical result sheets from participants' routine care. Such results routinely include glycated haemoglobin level (HbA1c) systolic/diastolic blood pressure, total cholesterol, low-density lipoprotein cholesterol (LDL), high density lipoproteins (HDL), and triglycerides. Any such information will be analysed and where appropriate help to address the research questions.

No restrictions will be placed on the care provided by healthcare professionals treating participants but use of prescribed and non-prescribed treatments will be recorded.

Members of the PEMF device group will be invited to qualitative on-line focus groups or interviews. Participants will also be asked to participate in focus groups to explore their experiences of using the PEMF device, including participants' perceptions on how the device could be improved, any perceived impact on their diabetes and quality of life, and any adverse effects. Focus groups were chosen as the data-gathering method of choice, as the interaction helps participants to explore and refine their own experiences and perspectives. Two members of the research team will jointly conduct each focus group. The focus groups will be directed by a topic guide. Topic guides will be updated throughout the study to incorporate emerging themes. Focus groups will take place 3 months after the initiation of the PEMF intervention. Up to 5 focus groups will take place with patients using the PEMF device. Focus groups will be audio-recorded and transcribed verbatim.

The PEMF devices will be delivered to the homes of participants and all measures involve self-reporting to be conducted at participants' own homes.

Project milestones:

Milestone 1: Pre-study preparation (2 months)

* produce study documents (information sheets, consent forms)
* obtain ethical approval

Milestone 2: Recruitment/ data collection (6 months)

* recruitment of 60 patients to the study
* obtain all baseline and follow-up outcome measures
* complete all focus groups
* mid-term report to study funders

Milestone 3: Data analysis (2 months)

* statistical analysis of data from outcome measures
* analysis of data from qualitative focus groups

Milestone 4: Dissemination

* end of study report to funders
* dissemination of findings to participants
* dissemination through conferences and peer reviewed journal articles

Data analysis-

Quantitative data- Appropriate descriptive statistics will be estimated for all baseline sociodemographic and clinical variables by arm, and for outcome variables (scores on). The association between baseline sociodemographic or clinical variables and outcome variables will be assessed using appropriate between-group tests or correlations depending on skewness. Primary outcome variables will be compared between the arms using t-tests, one-way analysis of variance, Mann-Whitney tests and Kruskal-Wallis tests, bearing in mind any skewness in the data. Data will also evaluate the impact of medication on outcome, comparing treatment outcomes from those on diabetic medication compared to those not currently receiving medication for their diabetes. An intention-to-treat analysis model will be followed.

Qualitative data- Data will be analysed inductively, using thematic analysis. One of the researchers will immerse themselves in the data, repeatedly reading the transcripts to understand participants' experiences. Key issues, concepts and themes arising from the data will be identified to create a coding framework. Transcripts will then be coded and analysed thematically.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years, of any gender.
* Consulted at their general practice for type 2 diabetes in the previous 12 months.
* Residing within England (due to delivery difficulties from covid-19).
* Self-reported confirmed diagnosis of type 2 diabetes.
* Self-reported stable medication regime for diabetes for at least one month.
* Sufficient command of English to complete questionnaires.
* Patients willing to participate in the study and be randomised into one of the two study groups.

Exclusion Criteria:

* Patients with type 1 diabetes.
* Patients with previous experience of using PEMF devices.
* Patients residing outside England.
* Patients with electronic implants such as pacemakers.
* Patients with an electro-cardio implant.
* Patients who have any electronic heart or lung apparatus.
* Patients who are pregnant.
* Patients who have a malignant tumour.
* Patients who are receiving high-level treatment.
* Patients who have a life-threatening illness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in score of the Appraisal of Diabetes Scale (ADS) | Baseline and at the end of the 3 months
  Appraisal of Diabetes Scale (ADS): The ADS is a brief 7-item patient-reported scale that assesses the impact of diabetes on a patient's life. The items, which were developed based on theory and previous research, include "How upsetting is having diabetes for you?" and "To what degree does your diabetes get in the way of your developing life goals?". The instrument has been shown to have acceptable internal consistency reliability, test-retest reliability, and construct validity. Higher scores indicate greater negative impact of diabetes.
Change in Measure Yourself Medical Outcome Profile (MYMOP)2 score | Baseline and at the end of the 3 months
  MYMOP2 is a validated questionnaire where patients can express their any two concerns and rate them
Change in the EQ-5D-5L tool score | Baseline and at the end of the 3 months
  EQ-5D-5L: Health related quality of life (HRQoL) will be measured using the EQ-5D-5L, which contains five indices to represent patients' HRQoL on the day of completing the form: mobility; self-care; usual activities; pain/discomfort; and anxiety/depression. The EQ-5D-5L also includes a visual analog scale (VAS), which records the respondent's self-rated health status on a graduated (0-100) scale, with higher scores for higher HRQoL. The EQ-5D-5L is well validated and numerous studies have used the EQ-5D-5L in a variety of patient populations, including diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Majumdar, Principal Investigator — St Marys University
Locations (1):
- St Marys University, Twickenham, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adu MD, Malabu UH, Malau-Aduli AEO, Malau-Aduli BS. Enablers and barriers to effective diabetes self-management: A multi-national investigation. PLoS One. 2019 Jun 5;14(6):e0217771. doi: 10.1371/journal.pone.0217771. eCollection 2019. PMID 31166971
- [Background] Chen L, Duan X, Xing F, Liu G, Gong M, Li L, Chen R, Xiang Z. Effects of pulsed electromagnetic field therapy on pain, stiffness and physical function in patients with knee osteoarthritis: A systematic review and meta-analysis of randomized controlled trials. J Rehabil Med. 2019 Dec 16;51(11):821-827. doi: 10.2340/16501977-2613. PMID 31583420
- [Background] Kaur S, Pandhi P, Dutta P. Painful diabetic neuropathy: an update. Ann Neurosci. 2011 Oct;18(4):168-75. doi: 10.5214/ans.0972-7531.1118409. PMID 25205950
- [Background] Paolucci T, Pezzi L, Centra AM, Giannandrea N, Bellomo RG, Saggini R. Electromagnetic Field Therapy: A Rehabilitative Perspective in the Management of Musculoskeletal Pain - A Systematic Review. J Pain Res. 2020 Jun 12;13:1385-1400. doi: 10.2147/JPR.S231778. eCollection 2020. PMID 32606905
- [Background] Relton C, Torgerson D, O'Cathain A, Nicholl J. Rethinking pragmatic randomised controlled trials: introducing the "cohort multiple randomised controlled trial" design. BMJ. 2010 Mar 19;340:c1066. doi: 10.1136/bmj.c1066. No abstract available. PMID 20304934
- [Background] Schwartz D, Lellouch J. Explanatory and pragmatic attitudes in therapeutical trials. J Clin Epidemiol. 2009 May;62(5):499-505. doi: 10.1016/j.jclinepi.2009.01.012. PMID 19348976
- [Background] Witt CM. Efficacy, effectiveness, pragmatic trials--guidance on terminology and the advantages of pragmatic trials. Forsch Komplementmed. 2009 Oct;16(5):292-4. doi: 10.1159/000234904. Epub 2009 Aug 25. No abstract available. PMID 19887807
- [Background] Yang X, He H, Ye W, Perry TA, He C. Effects of Pulsed Electromagnetic Field Therapy on Pain, Stiffness, Physical Function, and Quality of Life in Patients With Osteoarthritis: A Systematic Review and Meta-Analysis of Randomized Placebo-Controlled Trials. Phys Ther. 2020 Jul 19;100(7):1118-1131. doi: 10.1093/ptj/pzaa054. PMID 32251502